CLINICAL TRIAL: NCT01350518
Title: Dietary Intervention for Visceral Adiposity-Pilot
Brief Title: Dietary Intervention for Visceral Adiposity
Acronym: DIVA-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00013678
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: Intra-Abdominal Fat; Metabolic Syndrome; Hepatic steatosis
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study prepared meals and placebo (Placebo Comparator): Participants will have meals designed specifically for them based on their caloric needs. Participants will choose a weeks worth of meals (from a menu) and pick them up from the Clinical Research Unit twice a week. Participants will not receive any fiber (Benefiber) supplementation in their TrueLemon mixture.
  Interventions: Dietary Supplement: TrueLemon
- Nutritional Counseling with fiber (Active Comparator): Participants receiving nutritional education will have two individual sessions (spaced approx. 2 weeks apart). The nutritional sessions will focus on knowledge, self-regulation, motivation, experience and environment. Participants will receive fiber (Benefiber) supplementation as the fiber intervention in their TrueLemon mixture .
  Interventions: Dietary Supplement: Benefiber
- Nutrition counseling and placebo (Placebo Comparator): Participants receiving nutritional education will have two individual sessions (spaced approx. 2 weeks apart). The nutritional sessions (interventions) will focus on knowledge, self-regulation, motivation, experience and environment.Participants will receive no fiber supplementation in their TrueLemon mixture .
  Interventions: Dietary Supplement: TrueLemon
- Study prepared meals and fiber (Active Comparator): Participants will have meals designed specifically for them based on their caloric needs. Participants will choose a weeks worth of meals (from a menu) and pick them up from the Clinical Research Unit twice a week. Participants will receive fiber (Benefiber) supplementation as the fiber intervention in their TrueLemon mixture.
  Interventions: Dietary Supplement: Benefiber

INTERVENTIONS:
Dietary Supplement: Benefiber — Benefiber® powder will be used as our dietary supplement intervention. Benefiber® powder contains wheat dextrin, a 100% natural fiber. Participants in the intervention arm will receive 3 supplement packets to be consumed per day.
  Each active dietary supplement packet contains 8 grams of Benefiber® powder and 3 grams of TRUE® lemon flavoring, a 100% natural with no artificial ingredients or sweeteners, preservatives, sodium or gluten.
  Arms: Nutritional Counseling with fiber; Study prepared meals and fiber
Dietary Supplement: TrueLemon — Each placebo dietary supplement packet contains 8 grams of Splenda and 3 grams of TRUE® Lemon sweetener. Each packet is designed to be added to 8 oz of fluid. The three packets should be consumed each day in a total of 24 fluid ounces.
  Arms: Nutrition counseling and placebo; Study prepared meals and placebo

SUMMARY:
The purpose of this research study is to determine whether increased intake of dietary fiber during a 12-week, low-calorie weight loss intervention affects abdominal fat change and improves cardiovascular risk factors in African-American women more than a standard weight loss intervention.

The investigators are testing two main hypothesis:

Hypothesis 1: Women in the high dietary fiber intervention group will lose significantly more abdominal fat around their organs than women in the standard fiber group.

Hypothesis 2: Women in the high dietary fiber intervention group will have lower blood pressure, fasting glucose, fasting lipids and inflammatory factors at 3-months compared to women in the control group.

DETAILED DESCRIPTION:
OBJECTIVES:

Specific Aim 1: To test, in a small clinical trial of 30 pre-menopausal African American women, whether increased intake of dietary fiber embedded in a 12 week weight loss intervention will reduce VAT accumulation more than a standard weight loss intervention.

Hypothesis 1: Women in the high dietary fiber intervention group will lose significantly more VAT than women in the standard fiber group.

Specific Aim 2: To test, in a small clinical trial of 30 pre-menopausal African American women, whether increased intake of dietary fiber embedded in a 12 week weight loss intervention will improve cardiovascular risk factors more than a standard weight loss intervention.

Hypothesis 2: Women in the high dietary fiber intervention group will have lower blood pressure, fasting glucose, fasting lipids and inflammatory factors at 3-months compared to women in the control group.

Specific Aim 3: To characterize our ability to recruit and retain 30 African-American, premenopausal women to a 12 week weight loss intervention study

Specific Aim 4: To determine participant compliance with serum and other measurement evaluations and dietary compliance logs.

METHODS AND MEASURES

Design:

This study will be a randomized masked controlled trial design of 30 pre-menopausal African American women aged 20-50 years with BMI ≥ 30 kg/ m2 and waist circumference > 88 cm evaluating the effect of fiber supplementation on change in abdominal fat deposition. The fiber intervention will be nested within a 3-month weight loss trial. The placebo and active interventions will appear identical to the participant. The only person who will know of the intervention (fiber vs. placebo) is the Clinical Research Unit (CRU) (former General Clinical Research Center) Nutrition staff. All women will have ~ 800 kcal/day calorie restriction, for 12 weeks, designed lead to 0.5 kg - 0.9 kg per wk weight loss or 9-18 kg lost during the study. Diets will all contain at least 0.8 grams of protein/kg IBW and be limited to 15 grams total fiber. Calorie restriction will occur either through CRU prepared meal replacements or participant instituted calorie restriction learned via nutritional education sessions. Participants will be randomized and started on the 12-week study intervention on a rolling basis. At any one time, there will be 8 women enrolled in the study. The enrollment will continue until all 30 women are started. The women will not be held and then started as a group.

Randomization:

Although enrollment will be rolling, participants will be randomized in groups of eight to ensure that the capacity of the metabolic kitchen is always maintained. The randomization will be to one of four groups (1- intervention/feeding; 2- intervention/nutritional education; 3- placebo/feeding; 4-placebo/nutritional education). Participants will be randomized to one of these four groups at the close of her baseline visit. Randomization will occur via envelope. There will be an envelope for fiber intervention and one for caloric restriction method. The intervention envelope will contain four fiber cards (marked B) and four placebo cards (marked A). The calorie restriction envelope will contain for meal replacement cards (marked D) and four nutrition education cards (marked C). Participants will be given randomization assignment by CRU staff. The PI and participants will be blinded to the fiber intervention.

Setting:

This study will take place in two main settings, the CRU and each participant's home. All clinical measurements, nutritional education, meal replacement pick- up and distribution dietary supplements will take place at the CRU. The CRU has agreed to: 1) perform CT, RMR, and anthropomorphic measures as indicated for screening, baseline and 12-week follow-up; 2) draw, process and assay blood, as indicated, for screening, baseline and 12-week follow-up; 2) to provide two nutritional education sessions, two weeks apart (for the nutrition education group); 3) to prepare and distribute lunch and dinner (for the meal replacement group); 4) prepare and distribute daily fiber supplements for all participants; and 5) to prepare, distribute and collect weekly food compliance logs from each participant.

Interventions:

Dietary Fiber Intervention:

Benefiber® powder will be used as our dietary supplement intervention. Benefiber® powder contains wheat dextrin, a 100% natural fiber. It's taste-free, sugar-free, dissolves completely in noncarbonated beverages and soft foods, and won't thicken. Benefiber® powder can be mixed into any hot or cold beverage such as water, coffee, or juice; into soft foods such as applesauce, pudding or yogurt; or cooked into recipes for such foods as muffins, sauces or soups, without affecting the taste or consistency. Benefiber® powder is not recommended for carbonated beverages. Benefiber has a shelf life of 2 years when stored at a controlled room temperature of 20-25°C (68-77°F). Benefiber® Powder, which contains less than 20 ppm of gluten and is therefore considered "gluten-free," based on both the FDA and the Codex Alimentarius Commission's proposed definition of less than 20 ppm. Participants in the intervention arm will receive 3 supplement packets to be consumed per day.

Each active dietary supplement packet contains 8 grams of Benefiber® powder and 3 grams of TRUE® lemon flavoring, a 100% natural with no artificial ingredients or sweeteners, preservatives, sodium or gluten. The TRUE® Lemon product is made from cold-pressed and crystallized lemons which contain 0 calories and 0g carbohydrates. Each placebo dietary supplement packet contains 8 grams of Splenda and 3 grams of true lemon sweetener. Each packet is designed to be added to 8 oz of fluid. The three packets should be consumed each day in a total of 24 fluid ounces.

Weight Loss Methods:

All participants will have a daily caloric restriction of ~ 800 kcal in order to facilitate a loss of 0.5 kg - 0.9 kg per week weight loss or a 9-18 kg loss during the 12-week study period. All participants will undergo a resting metabolic rate determination using MedGraphics Ultima™ metabolic cart and the accompanying Breeze software. Based on the caloric need determined to maintain weight, a new caloric plan, 800 kcal lower than basal needs, will be determined. At minimum, however, all women will receive 1000 kcal per day. Once caloric goals are determined, these will be achieved with through CRU-prepared meal replacements or participant- instituted calorie restriction techniques learned via nutritional education group sessions.

Participants receiving nutritional education will two individual sessions (spaced approx. 2 weeks apart). The nutritional sessions will focus on knowledge, self-regulation, motivation, experience and environment.

All participants will be weighed at baseline and then weekly until the close of the study, week 13. Additionally, all participants will, with CRU-prepared meals, be asked to return uneaten food, record any foods eaten that were not part of the plan and complete weekly food compliance logs. Participants with self-directed food selection after nutritional education will be asked to completed detailed records of foods selected each day. All logs and food records will be reviewed by the PI and the CRU study dietician. If participants have: 1) increased weight by ≥ 5 pounds between weigh-in sessions; 2) a trend of weight gain for two consecutive sessions; or 3) failed to return 2 consecutive food logs; they will be flagged for additional nutritional counseling.

OUTCOMES Study Outcomes: The primary outcome, change in VAT between baseline and 12 weeks, will be obtained via repeat computed tomography (CT) scans. The secondary outcomes are change in CVD risk factors (blood pressure, fasting lipids, insulin sensitivity, C-reactive protein) and liver attenuation. Abdominal fat mass will be measured at the L4/L5 vertebral regions by CT. Height and weight will be measured to the nearest 0.5 cm and 0.1 kg, respectively, and BMI will be calculated (kg/m2). Systolic and diastolic blood pressure will be obtained after a 5-minute rest; the average of the final two of three measurements will be used in analysis. Fasting blood samples will be collected for the measurement of glucose, insulin, LDL, HDL,25-OH vitamin D, ghrelin, adiponectin, TNF-alpha, IL-6 and high sensitivity C-reactive protein. Insulin resistance will be calculated via a HOMA model. Covariates such as smoking status, physical activity, alcohol intake, sleep, and depressive symptoms will be ascertained at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal
* Self-identified as an African-American woman
* Aged 20-50 years
* Willing and able to provide informed consent
* No contraindication to weight loss

Exclusion Criteria:

* Diabetes or currently taking medication to lower blood sugar
* Currently on lipid lowering medications
* Currently taking chronic steroids
* Current diagnosis of kidney or heart failure
* Untreated hypothyroidism or hyperthyroidism
* BMI < 30 kg/m2 or waist circumference < 88 cm
* Current fiber supplementation
* Current pregnancy
* Body mass > 140 kg (CT limit)
* Inability to speak or read English
* Gastrointestinal disorders that prohibit the increased consumption of fiber
* Current participation in a structured weight loss/diet intervention program
* Inability to consume artificial sweeteners
* Inability or unwillingness to travel to the CRU during operating hours at the required frequency.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in abdominal adiposity measured by CT | 12 weeks
  Change in area of three abdominal fat depots,namely visceral,subcutaneous and liver fat.

SECONDARY OUTCOMES:
Change in metabolic risk factors | 12 weeks
  glucose, insulin, lipids, inflammatory markers, adipokines, blood pressure, BMI, 25-OH vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Kristen G Hairston, MD MPH, Principal Investigator — Wake Forest Unversity Health Sciences
Locations (1):
- Wake Forest University Clinical Research Unit, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hairston KG, Scherzinger A, Foy C, Hanley AJ, McCorkle O, Haffner S, Norris JM, Bryer-Ash M, Wagenknecht LE. Five-year change in visceral adipose tissue quantity in a minority cohort: the Insulin Resistance Atherosclerosis Study (IRAS) family study. Diabetes Care. 2009 Aug;32(8):1553-5. doi: 10.2337/dc09-0336. Epub 2009 Jun 1. PMID 19487643
- [Background] Hairston KG, Bryer-Ash M, Norris JM, Haffner S, Bowden DW, Wagenknecht LE. Sleep duration and five-year abdominal fat accumulation in a minority cohort: the IRAS family study. Sleep. 2010 Mar;33(3):289-95. doi: 10.1093/sleep/33.3.289. PMID 20337186
- [Background] Liu J, Fox CS, Hickson DA, May WD, Hairston KG, Carr JJ, Taylor HA. Impact of abdominal visceral and subcutaneous adipose tissue on cardiometabolic risk factors: the Jackson Heart Study. J Clin Endocrinol Metab. 2010 Dec;95(12):5419-26. doi: 10.1210/jc.2010-1378. Epub 2010 Sep 15. PMID 20843952